CLINICAL TRIAL: NCT03262337
Title: An Observational Study Using a Smartphone-app Supported Electronic Survey and Localization Tracking to Map Risk Behaviors and Symptoms of Swiss Travelers to Thailand, China, India, Brazil, Peru and Tanzania From 2 Swiss Travel Clinics
Brief Title: TOURIST 2: Tracking Of Urgent Risks In Swiss Travelers
Acronym: TOURIST2
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2017_00412
Record Dates: First submitted 2017-08-16; First posted 2017-08-25 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2017-10

CONDITIONS: Travel Health; Mobile Health Technology (mHealth); Elderly Travelers; Chronic Diseased Travelers; Risk Behavior
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Elderly Travelers: approximately 135 travelers with an age >= 60 years will be enrolled
  Interventions: Other: none, this is an observational study
- Chronic diseased travelers: approximately 225 travelers with a chronic disease will be enrolled
  Interventions: Other: none, this is an observational study
- Healthy travelers: approximately 640 healthy travelers with be enrolled
  Interventions: Other: none, this is an observational study

INTERVENTIONS:
Other: none, this is an observational study — none, this is an observational study

SUMMARY:
New mobile Health (mHealth) technology creates an opportunity to approach travel medicine research in a different way, revolutionising our understanding of risks to travellers. Using mHealth technology, the Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich (UZH), developed a TRAVEL app in collaboration with the Eidgnössische Technische Hochschule (ETH) Zurich.

By using this new technology, an extensive collection of data (prospective collection of individual travel behaviour and experienced health events, mapping the travel itinerary via global positioning system (GPS), linking to publicly available local weather data and data on disease endemicity) can be combined and an unprecedented abundance of information on travel behaviour and experienced risks can be obtained. These data will allow a much better understanding of travel risk profiles using cluster analysis. By simultaneously recording health outcomes, the relationship between travel risk profiles and health events can be assessed. In this study, the investigators will address several major shortcomings in travel health in tropical and subtropical destinations by improving the understanding of poorly assessed and potentially underestimated health threats (e.g. risk of accidents and injury, mental health disorders), and travel risks specific to elderly travellers and travellers with chronic conditions. These findings will directly feed back into individual travel advice given by practitioners in Switzerland and finally world-wide.

DETAILED DESCRIPTION:
New mobile Health (mHealth) technology creates an opportunity to approach travel medicine research in a different way, revolutionising our understanding of risks to travellers. Using mHealth technology, the Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich (UZH), developed a TRAVEL app in collaboration with the Eidgnössische Technische Hochschule (ETH) Zurich.

By using this new technology, an extensive collection of data (prospective collection of individual travel behaviour and experienced health events, mapping the travel itinerary via global positioning system (GPS), linking to publicly available local weather data and data on disease endemicity) can be combined and an unprecedented abundance of information on travel behaviour and experienced risks can be obtained. These data will allow a much better understanding of travel risk profiles using cluster analysis. By simultaneously recording health outcomes, the relationship between travel risk profiles and health events can be assessed. In this study, the investigators will address several major shortcomings in travel health in tropical and subtropical destinations by improving the understanding of poorly assessed and potentially underestimated health threats (e.g. risk of accidents and injury, mental health disorders), and travel risks specific to elderly travellers and travellers with chronic conditions.

1000 clients traveling to Thailand, China, India, Brazil, Peru or Tanzania will be recruited from the Travel Clinics in Zurich and Basel and through advertising at local travel agents and the universities of ETH and UZH from September 2017 until February 2019. After completing an intake at the clinic, participants will be given the option to use their own Smartphone for data collection, or to use a phone owned by the UZH-EBPI during travel. Participants will use a data collection app for questionnaire responses during and after travel including: a daily questionnaire on travel behaviors, daily symptoms questionnaire, and localization tracking, showing the participants' travel path and locations.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Traveler to Thailand, China, India, Brazil, Peru or Tanzania
* German-speaking (level 3 or higher)
* Literate (able to read and write in German - level 3 or higher)
* Capable of operating Smartphone application for data collection
* Traveling to Thailand, China, India, Brazil, Peru or Tanzania for ≤ 4 weeks

Exclusion Criteria:

- not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study recruitment will be conducted at the University of Zurich Travel Clinic and the Travel Clinic at the Swiss Tropical and Public Health Institute.
  That means that individuals seeking pre-travel advice at one of the two Travel Clinics will be asked to participate based inclusion criteria defined above.
  Furthermore, patients with chronic diseases will be referred to the Travel Clinics by various specialized clinics at the University Hospitals of Zurich and Basel (Gastroenterology, Rheumatology, Pneumology, Cardiology)
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Self-reported risk behaviors | for a maximum of 4 weeks during travel
  The study participant will report on daily risk behaviors prior to, during and after travel in a daily app-based questionnaire

SECONDARY OUTCOMES:
Self-reported symptoms | for a maximum of 4 weeks during travel
  The study participant will report on experienced symptoms/health events prior to, during and after travel in a daily app-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Silja Bühler, Dr., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Andreas Neumayr, Basel, Canton of Basel-City
  - University of Zurich, Epidemiology, Biostatistics and Prevention Institute, Travel Clinic, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farnham A, Blanke U, Stone E, Puhan MA, Hatz C. Travel medicine and mHealth technology: a study using smartphones to collect health data during travel. J Travel Med. 2016 Sep 4;23(6):taw056. doi: 10.1093/jtm/taw056. Print 2016 Jun. PMID 27592821